CLINICAL TRIAL: NCT04333342
Title: Clinical Usefulness of Monitoring Heart Rate Using Wearable Devices in the Patients of Graves' Disease Who Discontinue Anti-thyroid Drugs
Brief Title: Heart Rate Monitoring by Wearable Devices in Graves' Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jae Hoon Moon, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B-1911/577/304
Record Dates: First submitted 2020-03-11; First posted 2020-04-03 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Graves' Disease in Remission (Disorder)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wearable device group (Experimental): Participants use wearable device and their heart rate and activity are monitored. If their resting heart rate (rHR) increase beyond the set range or they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If their rHR stay within set range and they have no symptoms and signs, they come to hospital and get tests for thyroid function 6 months after discontinuing anti-thyroid drugs.
  Interventions: Device: heart rate monitoring using wearable devices
- Control group 1 (No Intervention): articipants don't use wearable devices. If they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If they have no symptoms and signs, they come to hospital and get tests for thyroid function 6 months after discontinuing anti-thyroid drugs.
- Control group 2 (No Intervention): Participants don't use wearable devices. If they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If they have no symptoms and signs, they come to hospital and get tests for thyroid function 3 and 6 months after discontinuing anti-thyroid drugs.

INTERVENTIONS:
Device: heart rate monitoring using wearable devices — Using Fitbit (TM) wearable devices, heart rate, activity data are collected. Based on these data, resting heart rate is monitored daily basis. If resting heart rate increase beyond set range, users are notified to visit the hospital.
  Arms: Wearable device group

SUMMARY:
A multi center randomized controlled study including 3 arms (wearable device group, control group 1, control group 2). This study is to investigate clinical feasibility of heart rate monitoring using wearable devices to detect disease recurrence in the patients who discontinue anti-thyroid drugs in remission state.

DETAILED DESCRIPTION:
A multi center randomized controlled study including 3 arms (wearable device group, control group 1, control group 2).

Study participants: Patients with Graves' disease who are planned to discontinue anti-thyroid drugs in remission state Wearable device group: Participants use wearable device and their heart rate and activity are monitored. If their resting heart rate (rHR) increase beyond the set range or they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If their rHR stay within set range and they have no symptoms and signs, they come to hospital and get tests for thyroid function 6 months after discontinuing anti-thyroid drugs.

Control group 1: Participants don't use wearable devices. If they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If they have no symptoms and signs, they come to hospital and get tests for thyroid function 6 months after discontinuing anti-thyroid drugs.

Control group 2: Participants don't use wearable devices. If they have hyperthyroid symptoms and signs, they should come to the hospital and get tests for thyroid function. If they have no symptoms and signs, they come to hospital and get tests for thyroid function 3 and 6 months after discontinuing anti-thyroid drugs.

A period to detecting disease recurrence, thyroid function test and Hyperthyroid Symptom Scale (HSS) at the time of disease recurrence, and the number of hospital visit and medical cost until detecting disease recurrence will be compared among 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Graves' disease who are being treated with anti-thyroid drugs (ATDs) and planned to discontinue ATDs
* Those who have who have continued to administer ATDs for more than 1 year
* Those who showed normal findings on thyroid function tests while maintaining stable doses of ATDs in the last 3 months
* Those who can use wearable devices and smartphone apps to work with during the research period

Exclusion Criteria:

* Those with heart disease, such as arrhythmia, that can affect heart rate
* Those who are taking medications that may affect their heart rate
* Those who researchers deemed unsuitable for participation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The time period to detecting disease recurrence (days) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  The time period to detecting disease recurrence after discontinuing anti-thyroid drugs
free T4 levels (ng/dL) | baseline, at the date of randomization
  thyroid function test at the time of disease recurrence
free T4 levels (ng/dL) | 3 months
  thyroid function test at the time of disease recurrence
free T4 levels (ng/dL) | 6 months
  thyroid function test at the time of disease recurrence
free T4 levels (ng/dL) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  thyroid function test at the time of disease recurrence
TSH levels (mIU/L) | baseline, at the date of randomization
  thyroid function test at the time of disease recurrence
TSH levels (mIU/L) | 3 months
  thyroid function test at the time of disease recurrence
TSH levels (mIU/L) | 6 months
  thyroid function test at the time of disease recurrence
TSH levels (mIU/L) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  thyroid function test at the time of disease recurrence
Hyperthyroid Symptom Scale (HSS, points) | baseline, at the date of randomization
  Hyperthyroid Symptom Scale at the time of disease recurrence
Hyperthyroid Symptom Scale (HSS, points) | 3 months
  Hyperthyroid Symptom Scale at the time of disease recurrence
Hyperthyroid Symptom Scale (HSS, points) | 6 months
  Hyperthyroid Symptom Scale at the time of disease recurrence
Hyperthyroid Symptom Scale (HSS, points) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  Hyperthyroid Symptom Scale at the time of disease recurrence

SECONDARY OUTCOMES:
the number of hospital visit until detecting disease recurrence (visit) | 3 months
  the number of hospital visit until detecting disease recurrence after discontinuing anti-thyroid drugs
the number of hospital visit until detecting disease recurrence (visit) | 6 months
  the number of hospital visit until detecting disease recurrence after discontinuing anti-thyroid drugs
the number of hospital visit until detecting disease recurrence (visit) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  the number of hospital visit until detecting disease recurrence after discontinuing anti-thyroid drugs
medical cost until detecting disease recurrence (KRW and USD) | 3 months
  medical cost until detecting disease recurrence after discontinuing anti-thyroid drugs
medical cost until detecting disease recurrence (KRW and USD) | 6 months
  medical cost until detecting disease recurrence after discontinuing anti-thyroid drugs
medical cost until detecting disease recurrence (KRW and USD) | at the time of disease recurrence, from date of randomization until the date of first documented recurrence of Graves' disease by thyroid function test, assessed up to 180 days
  medical cost until detecting disease recurrence after discontinuing anti-thyroid drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Moon, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (6):
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Chung-Ang University Hospital, Seoul
  - Eulji University Nowon Eulji Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of privacy issues